CLINICAL TRIAL: NCT06722755
Title: Optimizing Adherence to the Treatment of Sleep Apnea Among Patients With Stroke Undergoing Inpatient Rehabilitation
Brief Title: Stroke and CPAP Outcome Study 3 Randomized Controlled Trial
Acronym: SCOUTS3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sandeep Khot, Professor, Department of Neurology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00021430; R01HL164394-01A1 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-12-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: Stroke Patients; CPAP; OSA - Obstructive Sleep Apnea
Keywords: behavioral therapy; continuous positive airway pressure; stroke recovery; self determination; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intensive Support (Experimental): The Intensive Support (IS) group will receive the multicomponent intensive behavioral adherence program, which includes a CPAP technical support intervention, Motivational Enhancement Therapy (MET), and a Mobile Health intervention. Participants assigned to the IS group will also receive the 3 basic supportive treatments, including OSA and CPAP education, respiratory therapy and nursing support during inpatient rehabilitation, and referral to a DME company after inpatient rehabilitation discharge if needed.
  Interventions: Device: CPAP device; Behavioral: CPAP technical support; Behavioral: Phone follow-up for adherence feedback and self-management skills; Behavioral: myAir; Behavioral: Tailored messages; Behavioral: Written Materials; Behavioral: Motivational Enhancement Therapy (MET)
- Standard Support (Active Comparator): Participants assigned to the control group will receive only the 3 basic supportive treatments, including OSA and CPAP education, respiratory therapy and nursing support during inpatient rehabilitation, and referral to a DME company after study completion if needed. CPAP will be set up by the respiratory therapist (or similar personnel) on the inpatient rehabilitation (IPR) unit with standard mask fitting and troubleshooting, if available. Assistance with mask placement will be provided by IPR nurses and respiratory therapy, as needed. The control interventions mimic usual care, which typically entails a setup by respiratory therapy and support for CPAP placement and device maintenance by IPR nurses.
  Interventions: Device: CPAP device

INTERVENTIONS:
Device: CPAP device — Eligible participants with OSA will be started on automatically-adjusting CPAP.
Behavioral: CPAP technical support — Trained personnel will conduct mask selection and fitting, provide continual troubleshooting, and train participants on CPAP.
  Arms: Intensive Support
Behavioral: Phone follow-up for adherence feedback and self-management skills — The research coordinator will call participants approximately monthly to provide any needed support.
  Arms: Intensive Support
Behavioral: myAir — Study personnel will assist participants in registering for and using the myAir (ResMed) self-tracking app. This app also provides a library of how-to videos and provides email updates to participants.
  Arms: Intensive Support
Behavioral: Tailored messages — Tailored text messages will be sent to participants. Two-way texting messaging will also be available between the study team and participants.
  Arms: Intensive Support
Behavioral: Written Materials — A binder of written educational materials will be provided to participants.
  Arms: Intensive Support
Behavioral: Motivational Enhancement Therapy (MET) — A trained sleep coach will conduct up to 5 MET sessions with participants and 2 sessions with a CPAP partner during the study time period.
  Arms: Intensive Support

SUMMARY:
The SCOUTS 3 study aims to test the effectiveness of an intensive CPAP (Continuous Positive Airway Pressure) therapy support program compared to usual care in stroke patients with obstructive sleep apnea (OSA) during inpatient rehabilitation (IPR).

The study is a multicenter randomized controlled trial (RCT) involving recruitment of about 250 participants across two institutions and randomization of about 200 participants. It compares an intensive support (IS) program for CPAP use with standard support (SS) to evaluate the effectiveness of the IS intervention in increasing CPAP usage during and after stroke rehabilitation. The Intensive Support (IS) group will receive a multicomponent intensive behavioral adherence program, which includes a CPAP technical support intervention, Motivational Enhancement Therapy (MET), and a Mobile Health intervention. Outcomes measured include CPAP adherence as measured by average nightly use in minutes between randomization and 3 months and the modified Rankin Scale (mRS-9Q) to evaluate stroke recovery.

DETAILED DESCRIPTION:
Within an investigator-initiated, phase 2 multicenter randomized controlled trial, we will test the effect of the multicomponent behavioral adherence intervention on 3-months of CPAP use among stroke patients with obstructive sleep apnea (OSA) and continuous positive airway pressure (CPAP) therapy initiated during inpatient rehabilitation (IPR). The study will be conducted at 2 IPR centers, University of Washington (UW) in Seattle, WA., and Rancho Los Amigos National Rehabilitation Center (RLANRC) in Los Angeles, CA. Over a ~3-year period, adult patients recovering from acute stroke within the past 30 days will be recruited upon IPR admission to these centers and tested for OSA through a simple, portable cardiorespiratory study with automated software. Eligible participants with OSA will be randomized to CPAP plus: either the adapted adherence intervention or control. All randomized subjects will be treated with auto-titrating CPAP or aCPAP. CPAP use will be measured electronically. Both groups will continue CPAP for a 3-month treatment period. We anticipate enrolling approximately 250 participants over the ~3 years of recruitment to randomize 200 eligible participants. The primary endpoint will be the average nightly minutes of CPAP use over the 90-day period, objectively measured, and the secondary outcome will be the Modified Rankin Scale-9 questions assessed at 3 months by phone.

ELIGIBILITY:
Inclusion criteria include:

1. Age 18 years or older
2. Head CT or brain MRI demonstrating an acute ischemic infarction or intraparenchymal hemorrhage within past 30 days
3. Person providing consent (patient or legally authorized representative (LAR)) able to be consented in English or Spanish.

Exclusion criteria include:

1. Unable to obtain informed consent from participant or LAR in English or Spanish
2. Incarcerated
3. Known pregnancy-determined by reviewing clinical data
4. Current mechanical ventilation, tracheostomy, or supplemental oxygen use > 4L/min
5. Use of positive airway pressure within 14 days prior to stroke
6. History of pneumothorax, bullous emphysema or other serious co-morbid conditions which limit CPAP use
7. Stroke related to tumors, vascular malformations or subarachnoid hemorrhage
8. Active use of sedative drugs that can interfere with testing for obstructive sleep apnea (OSA) including any benzodiazepine, barbiturate, general anesthesia, or conscious sedation within the prior 48 hours of the planned portable sleep apnea study
9. Anticipated inpatient rehabilitation length of stay < 5 nights
10. Co-morbid conditions that limit OSA testing or CPAP use in the judgement of the study team
11. Recent cranial or spinal surgery with known or possible CSF leak or pneumocephalus within past 3 months
12. Patients at significant risk of aspiration that could render the patient at risk of harm from use of CPAP, in the opinion of the site PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
CPAP Adherence | 3 months
  Average nightly minutes of CPAP use over the 90-day period is passively transmitted from a modem in each CPAP device via cellular service and securely accessed via the ResMed program, AirView. Alternatively, data cards can be obtained and downloaded.

SECONDARY OUTCOMES:
Stroke recovery measure | 3 months
  Functional disability (mRS-9Q) will be measured at ~90 days by phone [range 0-5; higher scores indicate lower level of function in neurological disease]

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Khot, MD, MPH, Principal Investigator — University of Washington; Devin Brown, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Rancho Research Institute, Downey, California
  - University of Washington - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No